CLINICAL TRIAL: NCT00819403
Title: The Effects of Ezetimibe/Simvastatin Versus Simvastatin Alone on Platelet and Inflammatory Biomarkers in Patients With the Metabolic Syndrome
Brief Title: Simvastatin With or Without Ezetimibe and Atherothrombotic Biomarker Assessment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Michael Miller, Dr., University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00040970; MSP-JV IISP #32031
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Metabolic Syndrome
Keywords: triglycerides; hypertension; low hdl; obesity
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Obesity | interventions — Simvastatin; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- simvastatin (Active Comparator): Simvastatin 40 mg daily
  Interventions: Drug: simvastatin
- simvastatin/ezetimibe (Active Comparator): Subjects will receive 6 weeks of ezetimibe/simvastatin 10/40 mg, after which atherothrombotic biomarker assessment will be studied.
  Interventions: Drug: ezetimibe/simvastatin

INTERVENTIONS:
Drug: simvastatin — Subjects will receive 6 weeks of simvastatin 40 mg, after which atherothrombotic biomarker assessment will be studied.
  Other Names: zocor
  Arms: simvastatin
Drug: ezetimibe/simvastatin — Subjects will receive 6 weeks of ezetimibe/simvastatin 10/40 mg, after which atherothrombotic biomarker assessment will be studied.
  Other Names: vytorin
  Arms: simvastatin/ezetimibe

SUMMARY:
To determine whether the combination of ezetimibe and simvastatin improves biomarkers of atherothrombosis compared to simvastatin alone in patients with the metabolic syndrome.

DETAILED DESCRIPTION:
1. To assess the ex vivo effects of ezetimibe/simvastatin (E/S) (Vytorin 10/40mg) and simvastatin (S) (Zocor 40mg) on platelet and inflammation biomarkers in patients with documented metabolic syndrome.
2. To compare platelet-related effects including PAR-1 receptor inhibition of E/S with those of the established anti-platelet agents including aspirin, clopidogrel, intravenous and oral glycoprotein IIb/IIIa inhibitors.
3. To determine whether the addition of ezetimibe will yield extra protection beyond lipid modulation in the reduction of inflammation and platelet activation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women greater than or equal to 21 years of age
2. Diagnosis of metabolic syndrome. We defined the presence of metabolic syndrome based on the US National Cholesterol Education Program's Adult Treatment Panel III guidelines. Specifically, metabolic syndrome will be diagnosed and documented when 3 of the following 5 characteristics will be present:

   * abdominal obesity, given as waist circumference for men > 102 cm, and for women > 88 cm
   * triglycerides > 150 mg/dL
   * HDL cholesterol < 40 mg/dL for men, and < 50 mg/dL for women
   * blood pressure > 130/85 mm Hg
   * fasting glucose > 100 mg/dL

Exclusion Criteria:

1. Patients will be excluded for a history of bleeding diathesis
2. drug or alcohol abuse
3. prothrombin time greater than 1.5 times control
4. platelet count < 100,000/mm3
5. hematocrit < 25%
6. creatinine > 4.0 mg/dl
7. surgery or angioplasty performed within 3 months or planned for the future
8. history of gastrointestinal or other bleeding
9. history of drug-induced disorders
10. trauma, cancer, rheumatic diseases, coronary artery disease or stroke
11. Patients participating in other investigational drug trials within one month of completion will be also excluded
12. Patients treated with intravenous platelet glycoprotein IIb/IIIa inhibitors or thienopyridines, within past 6 months
13. Patients treated with statins or aspirin within past four weeks

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MICHAEL MILLER, MD, Principal Investigator — University of Maryland, College Park; VICTOR L. Serebruany, MD, PhD, Study Director — President, HeartDrug Research LLC
Locations (3):
- United States (3):
  - VA Maryland Health Care System, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients have been recruited and 15 have successfully completed the study.
Pre-assignment Details: Patients excluded included those unable to tolerate statin and/or ezetimibe treatment
Groups:
- Simvastatin Then Simvastatin/Ezetimibe: Simvastatin 40 mg daily then simvastatin/ezetimibe 10/40 mg daily
  Subjects will receive 6 weeks of simvastatin 40 mg, after which atherothrombotic biomarker assessment will be studied. Subjects will then receive 6 weeks of simvastatin/ezetimibe 10/40 mg, after which atherothrombotic biomarker assessment will be studied.
- Simvastatin/Ezetimibe Then Simvastatin: Subjects will receive 6 weeks of simvastatin/ezetimibe 10/40 mg, after which atherothrombotic biomarker assessment will be studied. Subjects will then receive 6 weeks of simvastatin 40 mg, after which atherothrombotic biomarker assessment will be studied.
Period: First Intervention (6 Weeks)
Arm/Group | Simvastatin Then Simvastatin/Ezetimibe | Simvastatin/Ezetimibe Then Simvastatin
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | Simvastatin Then Simvastatin/Ezetimibe | Simvastatin/Ezetimibe Then Simvastatin
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Simvastatin Then Simvastatin/Ezetimibe | Simvastatin/Ezetimibe Then Simvastatin
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Simvastatin: Simvastatin 40 mg daily
  simvastatin : Subjects will receive 6 weeks of simvastatin 40 mg, after which atherothrombotic biomarker assessment will be studied.
- Simvastatin/Ezetimibe: Subjects will receive 6 weeks of ezetimibe/simvastatin 10/40 mg, after which atherothrombotic biomarker assessment will be studied.
  ezetimibe/simvastatin : Subjects will receive 6 weeks of simvastatin 40 mg, after which atherothrombotic biomarker assessment will be studied.
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Simvastatin/Ezetimibe | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (6.6) | 50.5 (12.6) | 48.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Ex Vivo Effects of Treatment With Vytorin Versus Zocor for 6 Weeks on Platelet Alpha Thrombin PAR-1 Receptor Expression
Description: Measured using whole blood flow cytometry
Time Frame: 6 weeks
Population: Based on power calculations
Measure: Mean (Standard Deviation); unit: ng/dl
Groups:
- Simvastatin: Simvastatin 40 mg daily for 6 weeks, after which atherothrombotic biomarker assessment will be studied.
- Simvastatin/Ezetimibe: Subjects will receive 6 weeks of ezetimibe/simvastatin 10/40 mg for 6 weeks, after which atherothrombotic biomarker assessment will be studied.
Arm/Group | Simvastatin | Simvastatin/Ezetimibe
Number analyzed (Participants) | 15 | 15
ng/dl
  PAR 1/4 antigen | 35.4 (5.2) | 34.5 (5.4)
  PAR 1/4 activity | 23.6 (4.3) | 22.5 (6.2)

2. Secondary Outcome: Biomarkers of Inflammation
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Simvastatin/Ezetimibe: Ezetimibe/simvastatin 10/40 mg daily for 6 weeks, after which atherothrombotic biomarker assessment will be studied.
Arm/Group | Simvastatin | Simvastatin/Ezetimibe
Number analyzed (Participants) | 15 | 15
mg/dl
  CRP | 3.51 (.48) | 3.57 (.34)
  IL-6 | 1.24 (.12) | 1.33 (.21)

ADVERSE EVENTS:
Arm/Group | Simvastatin | Simvastatin/Ezetimibe
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=15) | Simvastatin/Ezetimibe (N=15)
GI symptoms (Gastrointestinal disorders) | 2 (3) | 1 (1) — Gas, bloating, change in bowel movements
Muscle symptoms (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) — Aches, cramps
Fatigue (Psychiatric disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No